CLINICAL TRIAL: NCT05429788
Title: A Phase 1b/2a Randomized, Double-Blind, Placebo Controlled, Parallel Study to Evaluate the Safety, Tolerability, and Efficacy of Two Doses of RLS103 (CBD Technosphere® Inhalation Powder) in Subjects With Acute Anxiety Within Social Anxiety Disorder (SAD)
Brief Title: Safety, Tolerability, and Efficacy of RLS103 in Subjects With Acute Anxiety Within Social Anxiety Disorder (SAD)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Receptor Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC2022-01
Record Dates: First submitted 2022-06-14; First posted 2022-06-23 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose RLS103 (Experimental): 3 mg CBD inhaled dry powder
  Interventions: Drug: Low dose RLS103
- High dose RLS103 (Experimental): 6 mg CBD inhaled dry powder
  Interventions: Drug: High dose RLS103
- placebo (Experimental): placebo inhaled dry powder
  Interventions: Drug: placebo inhaled dry powder

INTERVENTIONS:
Drug: Low dose RLS103 — 3 mg CBD inhaled powder administered before public speaking challenge
  Arms: Low dose RLS103
Drug: High dose RLS103 — 6 mg CBD inhaled powder administered before public speaking challenge
  Arms: High dose RLS103
Drug: placebo inhaled dry powder — placebo inhaled powder administered before public speaking challenge
  Arms: placebo

SUMMARY:
This is a Phase 1b/2a clinical trial to evaluate the safety, tolerability, and efficacy of RLS103 (cannabidiol [CBD] inhaled dry powder) to relieve the anxiety induced by a public speaking challenge in adults with social anxiety disorder (SAD).

Subject participation will last 4 - 6 weeks. Upon signing an informed consent, all subjects will enter a screening phase lasting up to 3 weeks and including history, physical examination, laboratory tests, ECG, spirometry, and psychological tests. Subjects will undergo a public speaking test after screening tests are performed and eligibility is confirmed. One week after the completion of the public speaking test, subjects will come back for a follow-up visit that will involve a repeat of the safety and psychiatric assessments conducted during screening.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent form (ICF) indicating that they understand the purpose of the study and the procedures required for the study and are willing to participate in the study and attend all visits and requirements.
* Male or female 18 through 65 years of age, inclusive.
* Current diagnosis of SAD as defined in the MINI.
* Clinician-rated LSAS total score ≥75 at Screening (Visit 1).
* Clinician-rated Hamilton Depression Score 17-items total score <18 at Screening (Visit 1).
* Women of childbearing potential must commit to the consistent and correct use of an effective method of birth control throughout the study and must also have negative pregnancy test result at Screening (Visit 1), Baseline (Visit 2), and Visit 3. Effective methods of contraception include surgical sterilization of the subject, condoms with spermicide, diaphragm with spermicide, hormonal contraceptive agents (oral, transdermal, or injectable), or implantable contraceptive devices.
* Body mass index (BMI) between 18 and 32 kg/m2 (inclusive) with a body weight ≥50 kg.
* Non-smoker with no cigarettes, cigars, e-cigarettes, or nicotine-containing products used in the 1 month prior to Screening as confirmed by negative serum cotinine results (<10 ng/mL) at Screening.
* Negative viral serology test results (HIV-1/HIV-2, hepatitis B and C virus).
* Must have no medical contraindication to CBD, including known allergies or hypersensitivities to CBD or the excipients in RLS103.
* Must demonstrate the ability to use the inhaler correctly through a training tool and must be able to tolerate inhalation of a placebo powder.
* Must have the ability and willingness to attend the necessary clinic visits.

Exclusion Criteria:

* Any history of bipolar disorder (I or II), schizophrenia, schizoaffective disorder, psychosis, anorexia or bulimia, premenstrual dysphoric disorder, autism-spectrum disorder, or obsessive-compulsive disorder.
* Any other current Axis I disorder, other than SAD, which is the primary focus of treatment. Note that subjects with concurrent Generalized Anxiety Disorder are eligible for the study provided that Generalized Anxiety Disorder is not the primary diagnosis.
* Subject with alcohol or substance use disorder within the 1 year prior to study entry.
* In the opinion of the Investigator, has a significant risk for suicidal behavior during the course of their participation in the study, or
* At Screening (Visit 1): the subject scores "yes" on items 1 or 2 in the C-SSRS with reference to a 6-month period prior to Screening; or
* At Screening (Visit 1): the subject has had 1 or more suicidal attempts with reference to a 2-year period prior to Screening; or
* At Visit 2 or Visit 3: the subject scores "yes" on items 1 or 2 in the Suicidal Ideation section of the C-SSRS with reference to Screening; or
* The subject is considered to be an imminent danger to themself or others.
* Two or more documented failed treatment trials with a registered medication approved for SAD, in the last three years whereby an adequate treatment trial is defined as that described in the package insert for a particular drug during which the subject received an adequate medication dosage (defined as the treatment dose indicated in the package insert to obtain efficacy for that particular drug).
* Use of any psychotropic or beta blocker medications within 14 days before study entry (other than medication permitted for insomnia: eszopiclone, ramelteon, melatonin, zaleplon, zolpidem, or antihistamines).
* Use of any over-the-counter product, prescription product, or herbal preparation for treatment of the symptoms of anxiety or social anxiety within 30 days before study entry; concomitant use is prohibited during the study.
* Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the follow-up period.
* Currently using marijuana, marijuana cigarettes, cannabis-related products, or CBD; or have used any of these products within 3 weeks prior to Screening (at the discretion of the Investigator in consultation with the Sponsor, to be confirmed by a urine drug test at Screening).
* Any history of pulmonary disease, including bronchospastic respiratory disease (bronchial asthma), or chronic obstructive pulmonary disease.
* Clinically significant abnormal values for ECG, chest X-ray, or spirometry, or hematology, serum chemistry, or urinalysis at Screening as deemed appropriate by the Investigator, including:
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 × the ULN
* Total bilirubin >1.5 × ULN (isolated bilirubin >1.5 ×ULN is acceptable if total bilirubin and direct bilirubin <35%)
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Received an investigational medicinal product within 30 days or 5 half-lives prior to Baseline, whichever is longer.
* Donated blood or blood products or had substantial loss of blood (more than 500 mL) within 3 months before the first administration of study drug or intention to donate blood or blood products during the study.
* Fever (body temperature >38°C) or symptomatic viral or bacterial infection within 2 weeks prior to Screening, including confirmed active COVID-19.
* Had major surgery (general anesthetic) in the last 3 months or minor surgery (local anesthetic) in the last 1 month prior to Screening or have any pre-planned surgery or procedures that would interfere with the conduct of the study.
* Is an employee of the Investigator or study site, with direct involvement in the proposed study or other studies under the direction of that Investigator or study site, as well as family members of the employees or the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 1 week (visit 3 to follow up visit)
  Safety and tolerability of RLS103 will be assessed by evaluating the incidence and severity of treatment emergent serious adverse events (TESAEs), treatment emergent adverse events (TEAEs), and adverse events (AEs) leading to discontinuation from the study.

SECONDARY OUTCOMES:
Change in subject-reported anxiety | 1 week (Visit 2 to Visit 3)
  To evaluate and compare the average Subjective Units of Distress Scale (SUDS) between RLS103- and placebo-treated patients reported during the 5-minute performance phases of the Visit 2 and Visit 3 public speaking challenge
Change in CGI | 1 week (Visit 2 to Visit 3)
  Investigator's impression of improvement of anxiety via the Clinical Global Impressions Scale (CGI) from Visit 2 to Visit 3

OTHER OUTCOMES:
Changes in pulse rate in subjects with SAD | 10 minutes, assessed at Visit 2 and Visit 3
  Changes in physiologic measures of anxiety (pulse rate) from before and after the 5-minute performance phases of the public speaking challenges from Visit 2 to Visit 3
Changes in respiratory rate in subjects with SAD | 10 minutes, assessed at Visit 2 and Visit 3
  Changes in physiologic measures of anxiety (respiratory rate) from before and after the 5-minute performance phases of the public speaking challenges from Visit 2 to Visit 3
Changes in blood pressure in subjects with SAD | 10 minutes, assessed at Visit 2 and Visit 3
  Changes in physiologic measures of anxiety (blood pressure) from before and after the 5-minute performance phases of the public speaking challenges from Visit 2 to Visit 3

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Receptor 102, Los Angeles, California
  - Receptor 105, Oceanside, California
  - Receptor 103, Torrance, California

IPD SHARING:
Plan to Share IPD: No